CLINICAL TRIAL: NCT06987916
Title: A Single-Arm, Open-Label Clinical Study on the Efficacy and Safety of U01 (ssCART-19) in the Treatment of Relapsed or Refractory B-Cell Lymphoma
Brief Title: Efficacy and Safety Evaluation of U01(ssCART-19) in B-Cell Lymphoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai Tongji Hospital, Tongji University School of Medicine (Other)
Responsible Party: Principal Investigator, Wenjun Zhang, professor, Shanghai Tongji Hospital, Tongji University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: U01-01
Record Dates: First submitted 2025-05-15; First posted 2025-05-23 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: B Cell Lymphoma
Keywords: ssCART-19; Relapsed or Refractory B-Cell Lymphma; IL-6
MeSH Terms: conditions — Lymphoma, B-Cell; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ssCART-19 (Experimental): All enrolled patients in this arm will receive ssCART-19
  Interventions: Biological: ssCART-19

INTERVENTIONS:
Biological: ssCART-19 — autologous T cells transduced with a lentiviral vector containing anti-CD19 CAR and small hairpin RNA to silence the IL-6 gene
  Other Names: anti-CD19 CAR T with small hairpin RNA to silence the IL-6 gene

SUMMARY:
This is an open-label phase1 study to assess the safety and efficacy of U01(ssCART-19) cell therapy in the treatment of patients with refractory or recurrent B-cell lymphoma .

DETAILED DESCRIPTION:
Cytokine release syndrome (CRS) and immune effector cell-associated neurotoxicity syndrome (ICANS) are critical complications in CAR T-cell therapy. Research highlights IL-6 as a central driver of CRS, as activated CAR T-cells secrete this cytokine, which in turn stimulates monocytes to produce additional IL-6. To mitigate this risk, ssCART-19-a modified anti-CD19 CAR T-cell therapy-incorporates small hairpin RNA (shRNA) technology to silence the IL-6 gene, thereby reducing IL-6 secretion by both CAR T-cells and monocytes. This study aims to assess the safety and efficacy of the U01 (ssCART-19) therapy in patients with refractory or recurrent B-cell lymphoma .

ELIGIBILITY:
Inclusion Criteria:

1. Participants must voluntarily sign the informed consent form (ICF) and demonstrate good compliance.
2. Participants must meet the following requirements:

   1. Age ≥2 years and ≤75 years at the time of signing the ICF (both sexes eligible). For minors (<18 years), the legal guardian must sign after full disclosure; minors with decision-making capacity must co-sign with their guardians.
   2. Confirmed diagnosis of B-cell lymphoma according to the NCCN Clinical Practice Guidelines for B-Cell Lymphomas (3rd Edition, 2024) .
   3. Prior treatment requirements :

   Failure to achieve partial response (PR) after first-line therapy, or relapse within 12 months post-first-line therapy; Relapsed/refractory B-cell lymphoma after second-line therapy (one standard chemotherapy regimen + one salvage regimen).

   Prior treatments must include CD20 monoclonal antibody (unless CD20-negative tumor confirmed by the investigator) and anthracycline-based regimens .

   Additionally, meet one of the following:

   i. Ineligible for autologous stem cell transplantation (ASCT); ii. Refusal of ASCT; iii. Post-ASCT relapse. d) Refractory/relapsed status at screening: Relapse: Disease progression (PD) after achieving PR or complete response (CR);

   Refractory:

   i. No response to last-line therapy (PD during/after treatment, or stable disease [SD] lasting <6 months); ii. Post-ASCT relapse/PD (biopsy-confirmed), including relapse/PD within 12 months post-ASCT with SD/PD after salvage therapy2.
3. CD19 positivity confirmed by immunohistochemistry (IHC) of tumor tissue (preferably within 6 months).
4. At least one measurable lesion assessed by the Lugano Lymphoma Response Criteria (Cheson 2014) .
5. ECOG performance status score 0-3 .
6. Adequate bone marrow reserve at screening:

   Absolute lymphocyte count (ALC) ≥0.3×10⁹/L ; Platelet count (PLT) ≥30×10⁹/L .
7. Adequate organ function:

   AST/ALT ≤3×ULN (≤5×ULN if due to tumor infiltration); Total bilirubin ≤2×ULN (≤3×ULN for Gilbert syndrome with direct bilirubin ≤1.5×ULN); Serum creatinine ≤1.5×ULN or creatinine clearance ≥60 mL/min (Cockcroft-Gault formula); Oxygen saturation >91% on room air (dyspnea grade ≤1); Left ventricular ejection fraction (LVEF) ≥50% ; INR ≤1.5×ULN and APTT ≤1.5×ULN .
8. Negative pregnancy test (blood/urine) within 7 days before CAR-T infusion for women of childbearing potential. All participants must agree to use effective contraception during the study and for ≥1 year post-treatment.
9. Adequate venous access for leukapheresis or blood collection, with no contraindications to leukapheresis.
10. Expected survival ≥3 months .

Exclusion Criteria:

1. Concurrent malignancies , except for:

   Malignancies with disease-free survival (DFS) >3 years ; Carcinoma in situ ;
2. Active viral infections :

   Hepatitis B : Positive for HBe-Ab and/or HBc-Ab with HBV-DNA > lower limit of quantitation (LLOQ) ; Hepatitis C : Positive HCV-Ab with HCV-RNA > LLOQ ; Positive Treponema pallidum antibody (TP-Ab); Positive HIV antibody ;
3. Uncontrolled infections (bacterial, fungal, viral, mycoplasmal, or others) as determined by the investigator;
4. Clinically significant CNS diseases (current or history), including:

   Epilepsy, cerebrovascular ischemia/hemorrhage, dementia, cerebellar disorders, or CNS-related autoimmune diseases , deemed uncontrolled by the investigator;
5. Cardiovascular exclusion criteria :

   Cardiac angioplasty/stent placement within 12 months prior to signing ICF ; NYHA Class II-IV congestive heart failure , myocardial infarction, unstable angina, or other clinically significant cardiac history; QTe interval ≥480 ms (Fridericia correction) or LVEF <50% at screening;
6. Primary immunodeficiency ;
7. Severe immediate hypersensitivity to any study drug;
8. Live vaccine administration within 6 weeks prior to screening ;
9. Pregnancy or lactation ;
10. Active autoimmune diseases ;
11. Participation in another interventional clinical trial within 30 days prior to ICF signing ;
12. Other conditions deemed ineligible by the investigator.

Ages: 2 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-04-22 (Actual); Primary Completion 2028-04-22 (Estimated); Study Completion 2030-04-22 (Estimated)

PRIMARY OUTCOMES:
The types, frequency, and severity of treatment related adverse events | Day1 to Week 4
  After CAR-T cell infusion, we will observe the potential adverse events, especially Cytokine Release Syndrome(CRS) and neurotoxicity Using NCI Common Terminology Criteria for Adverse Events(CTCAE) V5.0
Objective response rate(ORR) | At 1,3,6,9,12,18 and 24 months post-treatment follow up
Duration of response (DOR) | At 1,3,6,9,12,18 and 24 months post-treatment follow up
Progression free survival(PFS) | At 1,3,6,9,12,18 and 24 months post-treatment follow up
Overall survival(OS) | At 1,3,6,9,12,18 and 24 months post-treatment follow up

SECONDARY OUTCOMES:
Kinetics of CAR-T cells | Day1 to Month 3
  Use flow cytometry or qPCR to monitor the kinetics of CAR-T cells
Monitoring changes in IL-6, ferritin, and CRP in peripheral blood following CAR-T cell infusion | Day1 to Month 3

CONTACTS AND LOCATIONS:
Overall Officials: Wenjun Zhang, Doctor, Principal Investigator — Tongji hospital of tongji university (Shanghai tongji hospital)
Locations (1):
- Shanghai Tongji Hospital ( Tongji Hospital of Tongji University), Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No